CLINICAL TRIAL: NCT06386341
Title: Quality of Life in Obstructive Sleep Apnea patiënts Treated With Maxillomandibular Advancement Surgery.
Brief Title: QoL in OSA patiënts Treated With MMA Surgery.
Acronym: QOMAS
Status: Recruiting | Type: Observational
Sponsor: Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: W23.154
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-08

CONDITIONS: Sleep Apnea, Obstructive; Quality of Life
Keywords: Sleep Apnea, Obstructive; Quality of Life; Surgery, Oral
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Patiënts who underwent MMA surgery for OSA.
  Interventions: Procedure: Maxillomandibular Advancement Surgery
- Control group: Patiënts who underwent MMA surgery for other reasons than OSA.
  Interventions: Procedure: Maxillomandibular Advancement Surgery

INTERVENTIONS:
Procedure: Maxillomandibular Advancement Surgery — Surgery where the upper and lower jaw are repositioned.

SUMMARY:
The aim of this observational study is to evaluate the impact of maxillomandibular advancement surgery on the quality of life in patients treated with obstructive sleep apnea.

The main question it aims to answer is:

Does MMA surgery in OSA patiënts improve their quality of life?

Patients will answer online surverys about their QoL and there will be data collected like length, weight and blood pressure.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact of MMA surgery on the quality of life of patients with obstructive sleep apnea.

It was hypnotized that MMA does not result in a significant improvement in the quality of life in patients with OSA.

The main objective is the SF-36 questionnaire The secondary objectives are the; OHIP-14, ESS, FOSQ, EQ-5D-3L and OQLQ

Design: observational study

Study population: 80 Patients who qualify for MMA above the age of 18

The patients will be recruited at the departments of Oral and Maxillofacial surgery. Individuals who match the next inclusion and exclusion criteria will be the population base of this study.There will also be a control group.These patients will have the same inclusion and exclusion criteria next to the diagnosis with OSA. The control group will be a group of patients without OSA.

Inclusion criteria for this research are:

* 18 years and older.
* Ability to speak, read and write Dutch.
* Ability to follow up.
* Ability to use a mobile device with internet connection for the online questionnaires.
* Diagnosis with OSA. (only for the intervention group)
* Expected to maintain current lifestyle (sports, medicine, diet etc.).
* Qualifies for MMA surgery
* Patients who provide informed consent

Exclusion criteria for this research:

* Patients who do not qualify for MMA surgery
* Medication used/ related to sleeping disorders.
* Night or shifting work.
* Severe chronic heart failure.
* Medical history of known causes of tiredness by day or severe sleep disruption (insomnia,
* PLMS, Narcolepsy).
* Seizure disorder.
* Known medical history of mental retardation, memory disorders or psychiatric disorders.
* Patients with old type of pacemakers (It is possible that old types of peacemakers are not
* Compatible with the electromagnetic radiation of the electronics of the SPT).
* Shoulder, neck and back complaints.
* Reversible morphological upper airway abnormalities (e.g. enlarged tonsils).
* Inability to provide informed consent.
* Simultaneous use of other treatment modalities to treat OSA.
* Previous treatment for OSA with MRA or SPT
* Pregnancy.
* patients under the age of 18
* Patients with mild or no OSA at all (if patient meets this criteria they will be part of the control group)

In total there will be 80 patients included.

There will be no intervention done for the purpose of this study. But the intervention that will be observed is how the MMA effects the Quality of Life of the patients who underwent this surgery. We are going to prospective observe them and follow them up through their procedure.

The responsible researcher will introduce the research to the patients. When patients meet the inclusion criteria they will be asked to participate in the research. The decision regarding participation in the study, which is made by the patient, is entirely voluntary. Patients are given two weeks time to consider joining the study population. Refusal of participation will have no consequences for further treatment of the patient. They will be asked to sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Ability to speak, read and write Dutch.
* Ability to follow up.
* Ability to use a computer with internet connection and windows-software for uploading data
* and online questionnaires.
* Diagnosis with OSA. (only for the intervention group)
* Expected to maintain current lifestyle (sports, medicine, diet etc.).
* Qualifies for MMA surgery
* Patients who provide informed consent

Exclusion Criteria:

* Patients who do not qualify for MMA surgery
* Medication used/ related to sleeping disorders.
* Night or shifting work.
* Severe chronic heart failure.
* Medical history of known causes of tiredness by day or severe sleep disruption (insomnia,
* PLMS, Narcolepsy).
* Seizure disorder.
* Known medical history of mental retardation, memory disorders or psychiatric disorders.
* Patients with old type of pacemakers (It is possible that old types of peacemakers are not
* Compatible with the electromagnetic radiation of the electronics of the SPT).
* Shoulder, neck and back complaints.
* Reversible morphological upper airway abnormalities (e.g. enlarged tonsils).
* Inability to provide informed consent.
* Simultaneous use of other treatment modalities to treat OSA.
* Previous treatment for OSA with MRA or SPT
* Pregnancy.
* patients under the age of 18
* Patients with mild or no OSA at all

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing maxillomandibular advancement surgery for OSA (intervention group) or other reasons (control group).
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
SF-36 | 5 minutes
  Survey

SECONDARY OUTCOMES:
OHIP-14 | 5 minutes
  Survey
ESS | 5 minutes
  Survey
FOSQ | 5 minutes
  Survey
EQ-5D-3L | 5 minutes
  Survey
OQLQ | 5 minutes
  Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonessenhuis, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No